CLINICAL TRIAL: NCT06125418
Title: Effect of Customized Healing Abutments on Peri-implant Soft Tissue and Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pimduen Rungsiyakull, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43/2022
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Peri-implant Tissue Response With Use of Customized Healing Abutments
Keywords: dental implant, customized healing abutment

STUDY DESIGN:
Intervention Model Description: patients in each group will received different types of customized healing abutment
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized group (Experimental): patients who received customized healing abutments following implant placement. customized healing abutments will be fabricated with different macrogeometry and different emergence angle
  Interventions: Procedure: customized healing abutment
- Standard group (Experimental): patients who received standard titanium healing abutments following implant placement
  Interventions: Procedure: standard healing abutment

INTERVENTIONS:
Procedure: customized healing abutment — patients will undergoes one-stage implant placement with customized healing abutments with different macrogeometry and emergence angle made prior to the surgery and will be inserted without sutures, after osseointegration completed patients will received single crown on implant.
  Arms: Customized group
Procedure: standard healing abutment — patients will undergoes one-stage implant placement with standard titanium healing abutment made prior to the surgery and will be inserted without sutures, after osseointegration completed patients will received single crown on implant.
  Arms: Standard group

SUMMARY:
The goal of this clinical trial is to evaluate effect of customized healing abutment in patients who need single implant reconstruction. The main question it aims to answer is:

• effect of customized healing abutment on peri-implant soft and hard tissue Participants will received customized healing abutments before final prostheses delivery.

DETAILED DESCRIPTION:
Patients who need single implant restoration will be received one- stage implant placement with utilization of customized healing abutment. Data collection about change in hard and soft tissue will be collected digitally at several times points. Patients will received single crown on implant as final prosthesis. Change in peri-implant tissue will be analyzed with digital softwares.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* patients who needed a single implant placing therapy in maxillary or mandibular arch except in third molar regions
* sufficient mesial distal and interocclusal space for placement of the implant and definitive restoration;
* had sufficient apical bone to place an implant with minimum primary stability of 30 Ncm.

Exclusion Criteria:

* medical and general contraindications for the surgical procedure;
* heavy smokers (>10 cigarettes/day);
* an active infection at the implant site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
soft tissue alteration | T0 baseline before implant placement,T1 1month follow up, 4month follow up, 6month follow up, 12month follow up
  peri-implant soft tissue change compared to baseline including vertical and horizontal soft tissue alteration by superimposing intraoral scan at different time points
hard tissue alteration | T0 baseline before implant placement, 6month follow up, 12month follow up
  peri-implant marginal bone change compared to baseline at different time points by periapical radiograph
volumetric alteration | T0 baseline before implant placement,T1 1month follow up, 4month follow up, 6month follow up, 12month follow up
  peri-implant volumetric change at different time points compared to baseline with superimposing intraoral scan

SECONDARY OUTCOMES:
pain numerical rating scale | at prosthesis delivery, 2 hours and 24 hours after prosthesis delivery
  pain assessment at time of final prosthesis delivery with scale from 0 to 10
pink esthetic score | T0 baseline before implant placement, 6 month follow up
  pink esthetic score change compared to before implant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pimduen Rungsiyakull, AssocProfDr, Principal Investigator — Chiang Mai University
Locations (1):
- Department of Prosthodontics, Faculty of Dentistry, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No